CLINICAL TRIAL: NCT07210723
Title: A Phase 2b/3, Adaptive, Randomized, Double-blind, Placebo-controlled, Multicenter Study to Assess the Efficacy and Safety of Danicamtiv in Participants With Symptomatic Genetic and Familial Dilated Cardiomyopathy
Brief Title: A Study of the Efficacy and Safety of Danicamtiv in Participants With Symptomatic Genetic and Familial Dilated Cardiomyopathy
Acronym: KINSHIP-DCM
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kardigan, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAN-301
Record Dates: First submitted 2025-09-23; First posted 2025-10-07 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Symptomatic Genetic Dilated Cardiomyopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- danicamtiv (Experimental)
  Interventions: Drug: danicamtiv
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: danicamtiv — Danicamtiv will be administrated twice daily for up to 26 weeks
  Arms: danicamtiv
Drug: Placebo — Placebo will be administrated twice daily for up to 26 weeks
  Arms: placebo

SUMMARY:
The Sponsor is studying an investigational medication called danicamtiv to determine if it can help people with genetic and familial dilated cardiomyopathy (DCM). Investigational means that the safety and effectiveness of danicamtiv have not been established. Currently, there are no approved drugs that are designed specifically to treat genetic or familial DCM.

The purpose of this study is to evaluate how well danicamtiv works compared to a placebo (sugar pill that looks like danicamtiv pill but does not contain any danicamtiv) and see how safe it is for people with genetic and familial DCM. In DCM, the heart muscle weakens and enlarges, making it harder for the heart to pump blood; this can happen for different reasons. Some people have DCM because of a change in a gene (called genetic DCM). Others may have DCM that runs in their family, even if no specific gene change is found (called familial DCM).

The main goals of the study are:

* To assess the effect of danicamtiv on cardiac function using echocardiogram.
* To evaluate the impact of danicamtiv on exercise capacity
* To evaluate the safety and tolerability of danicamtiv

Participants will:

* Take danicamtiv or placebo every day for approximately 6 months
* Visit the clinic about 12 times for initial evaluation, checkups, tests and follow up

ELIGIBILITY:
Key Inclusion Criteria:

1. Has a diagnosis of DCM due to probable disease-causing variants of MYH7, TTN, or other identified genetic DCM variants, or with familial DCM
2. Has New York Heart Association (NYHA) Class II-IV at Screening with stable symptoms for ≥1 month.
3. Has at least mild left ventricular enlargement (LVE) and has adequate acoustic windows to enable accurate TTEs according to the Echocardiography Core Laboratory.
4. Has a LVEF of ≤45%.
5. Is on stable doses of maximally tolerated standard-of-care heart failure (HF) therapies reflecting current guidelines for at least 4 weeks prior to the first visit.
6. Has DCM not attributed to substance abuse, amyloidosis, sarcoidosis, or any other secondary form of cardiomyopathy per the Investigator.
7. Can perform an upright cardiopulmonary exercise training (CPET) with a peak oxygen uptake (pV̇O2) of 80% or less of predicted for a healthy individual and respiratory exchange ratio (RER) of ≥1.05

Key Exclusion Criteria:

1. Has heart failure with reduced ejection (HFrEF) caused primarily by ischemic heart disease, chronic valvulopathy, or another condition, as determined by the Investigator.
2. Recent (<90 days) clinically significant cardiac events, including acute coronary syndrome, hemodynamically significant epicardial coronary disease (per Investigator), coronary revascularization (percutaneous coronary intervention [PCI] or coronary artery bypass graft [CABG]), or hospitalization for heart failure/intravenous (IV) diuretic use.
3. Presence of disqualifying cardiac rhythms that might interfere with reliable echocardiographic measurements of left ventricle (LV) function, as determined by the Investigator including: (a) inadequately rate-controlled atrial fibrillation, (b) ectopic beats (atrial, junctional or ventricular) of sufficient frequency (e.g. > 10% of total beats) that the participant's cardiac rhythm is irregular potentially interfering with reliable echocardiographic measurements of LV function.
4. Unstable or untreated severe ventricular arrythmia (eg, ventricular tachycardia or ventricular fibrillation).
5. History of malignancy of any type within 5 years prior to Screening
6. Severe renal insufficiency (defined at the time of Screening as current estimated glomerular filtration rate [eGFR] <15 mL/min/1.73m2 by simplified Modification of Diet in Renal Disease equation [sMDRD]).
7. History or evidence of any other clinically significant disorder, condition, or disease that, in the opinion of the Investigator or Sponsor, would pose a risk to participant safety or interfere with the study evaluation
8. History of heart transplantation or anticipated heart transplantation in the next 6 months.
9. Ongoing or anticipated advanced cardiac interventions, including chronic IV inotropic therapy, planned cardiac resynchronization therapy (CRT) or major surgery, or current/anticipated ventricular assist device placement within 6 months
10. Clinically significant laboratory abnormalities at Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Part 1: Change from Baseline (Day 1) to Week 26 in left atrial function index in Cohort 1 | 26 weeks
Part 2: Change from Baseline (Day 1) to Week 26 in peak VO2 in Cohort 1 | 26 weeks

SECONDARY OUTCOMES:
Part 1: Change from Baseline (Day 1) to Week 26 in peak VO2 | 26 weeks
Part 1: Association between response in left ventricular global longitudinal strain and/or left atrial function index after 2 weeks of active treatment with placebo-adjusted Week 26 response in peak VO2 | 26 weeks
Part 1: Change from Baseline (Day 1) to Week 26 in left atrial function index in overall population | 26 weeks
Part 1 and 2: Change from Baseline (Day 1) to Week 26 in left ventricular ejection fraction | 26 weeks
Part 1 and 2: Change from Baseline (Day 1) to Week 26 in ventilatory efficiency | 26 weeks
Part 1 and 2: Change from Baseline (Day 1) to Week 26 in Kansas City Cardiomyopathy Questionnare (KCCQ-23) Clinical Summary Score | 26 weeks
  All scores are represented on a 0-to-100-point scale, where lower scores represent more severe symptoms and/or limitations and scores of 100 indicate no symptoms, no limitations, and excellent quality of life.
Part 1: Proportion of participants from Baseline (Day 1) to Week 26 who achieve at least a one-class improvement in New York Heart Association (NYHA) class | 26 weeks
  NYHA is a system used to categorize the severity of heart failure symptoms based on a patient's functional capacity, where 1 indicates no symptoms or limitations and 4 indicates symptoms present at rest.
Part 2: Change from Baseline (Day 1) to Week 26 in left atrial function index | 26 weeks
Part 2: Change from Baseline (Day 1) to Week 26 in peak VO2 in the responder subgroup | 26 weeks
Part 2: Change from Baseline (Day 1) to Week 26 in peak VO2 in overall population | 26 weeks
Part 1 and 2: Change from Baseline (Day 1) to Week 26 in left ventricular global longitudinal strain | 26 weeks
Part 1 and 2: Percent change from Baseline (Day 1) to Week 26 in NT-proBNP concentrations | 26 weeks
Part 1 and 2: Characterization of peak (Cmax) of danicamtiv | 20 weeks
Part 1 and 2: Characterization of trough (Cmin) plasma concentrations of danicamtiv | 20 weeks

OTHER OUTCOMES:
Part 1 and 2: Incidence and severity of treatment emergent adverse events, adverse events of special interest, serious adverse events and disease related events | 26 weeks
Incidence of abnormal findings in laboratory assessments, physical examinations, 12-lead ECGs, and vital signs | 26 weeks

CONTACTS AND LOCATIONS:
Locations (11):
- United States (9):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Cedars Sinai, Los Angeles, California
  - UCSF, San Francisco, California
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
- United Kingdom (2):
  - NHS Greater Glasgow and Clyde, Glasgow
  - Hammersmith Hospital, Imperial College of London, London

IPD SHARING:
Plan to Share IPD: No